CLINICAL TRIAL: NCT04387305
Title: Traumatic Injury Clinical Trial Evaluating Tranexamic Acid in Children (TIC-TOC): An Efficacy Study
Brief Title: Traumatic Injury Clinical Trial Evaluating Tranexamic Acid in Children: An Efficacy Study
Acronym: TIC-TOC
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Daniel Nishijima, MD, MAS (Other)
Collaborators: Pediatric Emergency Care Applied Research Network (Network)
Responsible Party: Sponsor-Investigator, Daniel Nishijima, MD, MAS, Associate Professor, University of California, Davis
Organization: University of California, Davis (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 128206
Record Dates: First submitted 2020-05-05; First posted 2020-05-13 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Brain Injuries, Traumatic; Wounds and Injury; Hemorrhage; Trauma Injury
Keywords: Tranexamic acid; Brain Injuries; Hemorrhage; Clinical Trial; Children; Pediatric; Trauma
MeSH Terms: conditions — Brain Injuries, Traumatic; Wounds and Injuries; Hemorrhage; Accidental Injuries; Brain Injuries | interventions — Tranexamic Acid

STUDY DESIGN:
Intervention Model Description: Bayesian adaptive response
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Tranexamic acid 15 mg/kg bolus (Experimental): Subjects will receive a 15 mg/kg bolus of tranexamic acid over 30 minutes followed by a 2 mg/kg/h infusion over 8 hours. This represents 31 mg/kg total dose of TXA.
  Interventions: Drug: Tranexamic acid injection
- Tranexamic acid 30 mg/kg bolus (Experimental): Subjects will receive a 30 mg/kg bolus of tranexamic acid over 30 minutes followed by a 4 mg/kg/h infusion over 8 hours. This represents 62 mg/kg total dose of TXA.
  Interventions: Drug: Tranexamic acid injection
- Tranexamic acid 45 mg/kg bolus (Experimental): Subjects will receive a 45 mg/kg bolus of tranexamic acid over 30 minutes followed by a 6 mg/kg/h infusion over 8 hours. This represents 91 mg/kg total dose of TXA. This dosing arm will only open if a dose-effect is determined based on accumulating data.
  Interventions: Drug: Tranexamic acid injection
- Placebo (Placebo Comparator): Subjects in the placebo group will receive a bolus dose of normal saline over 10 minutes followed by a normal saline infusion over 8 hours
  Interventions: Drug: Tranexamic acid injection

INTERVENTIONS:
Drug: Tranexamic acid injection — Active drug is provided to participants as described based on the TXA arm they are randomized to.

SUMMARY:
Trauma is the leading cause of death and disability in children in the United States. The objective of this study is to evaluate the benefits and harms of tranexamic acid (TXA; a drug that stops bleeding) in severely injured children with hemorrhagic brain and/or torso injuries. Using thromboelastography, we will measure baseline fibrinolysis to assess for treatment effects of TXA at different levels of fibrinolysis.

DETAILED DESCRIPTION:
The TIC-TOC efficacy trial is a multicenter, adaptive allocation, randomized controlled trial of children younger than 18 years with hemorrhagic injuries to the torso and/or brain to evaluate the efficacy of TXA on functional outcome as measured by the PedsQL. Children will be randomized to one of three arms: 1) TXA 15 mg/kg bolus over 30 minutes, followed by a 2 mg/kg/hr infusion over 8 hours), 2) TXA 30 mg/kg bolus over 30 minutes, followed by a 4 mg/kg/hr infusion over 8 hours), and 3) normal saline placebo. A third TXA dose (45 mg/kg bolus dose over 30 minutes, followed by a 6 mg/kg/hr infusion over 8 hours) may be added later in the trial if a dose effect based on accumulating data is noted. The trial will be conducted in the Pediatric Emergency Care Applied Research Network (PECARN) across 40 sites over 4 years of enrollment for a maximum sample size of 2000 patients.

A Bayesian adaptive randomization design will be used to evaluate the efficacy of TXA in children with hemorrhagic brain and/or torso injuries. Because different types of injury have different pathophysiology and potential response to TXA, three different injury strata will be evaluated: isolated hemorrhagic brain injury, isolated hemorrhagic torso injury, and both hemorrhagic brain and torso injuries. The efficacy of TXA will be analyzed across all enrolled children as well as across each type of injury.

The Bayesian adaptive trial design also efficiently evaluates the effectiveness of TXA across different TXA doses. The trial will randomize the first 500 patients to two doses of TXA and placebo at a fixed 1:1:1 ratio. Interim analyses will be conducted when 500, 750, 1000, 1250, 1500, and 1750 patients have been enrolled. At each interim analysis, randomization probabilities will be adjusted in order to preferentially allocate patients to better performing doses, while allocation to the placebo arm will stay fixed. The adaptive randomization will be based entirely on pre-planned rules using accumulating data. A Bayesian hierarchical model will be used to estimate the treatment effect for each of the injury types to be informed by the data accumulated from all injury types. At interim analyses, if a dose effect is noted towards the higher dose of TXA (30 mg/kg bolus then a 4 mg/kg/hr infusion) being more efficacious using pre-specified criteria, then a higher dose study arm (TXA 45 mg/kg bolus then a 6 mg/kg/hr infusion) will be opened later in the trial. If the dose response curve is flat, suggesting that TXA is ineffective, then futility stopping rules can end the trial early.

ELIGIBILITY:
Inclusion Criteria:

1. Less than 18 years old AND
2. Penetrating torso trauma, blunt torso trauma, or head trauma as defined below:
3. Penetrating Torso Trauma:

   a. Penetrating trauma to the chest, abdomen, neck, or pelvis with at least one of the following:
   * age-adjusted hypotension, or
   * age-adjusted tachycardia despite adequate resuscitation fluids, or
   * radiographic evidence of internal hemorrhage, or
   * clinician suspicion of ongoing internal hemorrhage
4. Blunt Torso Trauma:

   1. Clinician suspicion of hemorrhagic blunt torso injury and at least one of the following:

      * age-adjusted hypotension, or
      * age-adjusted tachycardia despite adequate resuscitation fluids
   2. Hemothorax on chest tube placement or imaging,
   3. Clinical suspicion of hemorrhagic blunt torso injury and Intraperitoneal fluid on abdominal ultrasonography (Focused Assessment with Sonography in Trauma),
   4. Intra-abdominal injury on CT with either contrast extravasation or more than trace intraperitoneal fluid,
   5. Pelvic fracture with contrast extravasation or hematoma on abdominal/pelvic CT scan with at least one of the following:

      * Age-adjusted hypotension, or
      * Age-adjusted tachycardia.
5. Head Trauma:

   1. Initial Glasgow Coma Scale (GCS) score 3 to 13 with associated intracranial hemorrhage on cranial CT scan (enroll after cranial CT scan)

Exclusion Criteria:

* Unable to administer study drug within 3 hours of traumatic event
* Known pregnancy
* Known ward of the state
* Cardiac arrest prior to randomization
* GCS score of 3 with bilateral unresponsive pupils
* Isolated subarachnoid hemorrhage, epidural hematoma, or diffuse axonal injury
* Known venous or arterial thrombosis
* Known bleeding/clotting disorders
* Known seizure disorders
* Known history of severe renal impairment
* Known allergy to TXA
* Unknown time of injury (includes suspected non-accidental trauma)
* Previous enrollment into the TIC-TOC trial
* Prior TXA for current injury
* Prior opt-out
* Non-English and non-Spanish speaking

Ages: 0 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2000 (Estimated)
Dates: Start 2026-10-01 (Estimated); Primary Completion 2031-03-31 (Estimated); Study Completion 2031-03-31 (Estimated)

PRIMARY OUTCOMES:
Pediatric Quality of Life Inventory (PedsQL) area under the curve | 1 week, 1 month, 3 months, and 6 months (as measured as an area under the curve)
  Neurocognitive functioning and quality-of-life measure; 0 to 100 with higher scores representing better outcomes

SECONDARY OUTCOMES:
Intracranial hemorrhage progression | 24 hours (±6 hours)
  Intracranial hemorrhage progression on cranial computed tomography imaging
Blood transfusion | First 48 hours after randomization
  Total volume of packed red blood cells, platelets, fresh frozen plasma, and cryoprecipitate
PedsQL Physical Domain area under the curve | 1 week, 1 month, 3 months, and 6 months
  Physical domain of the PedsQL measure; 0 to 100 with higher scores representing better outcomes

OTHER OUTCOMES:
Glasgow Outcome Scale-Extended (GOS-E) Peds | 1 week, 1 month, 3 months, and 6 months
  Global functioning as measured on an 8-point scale (8-death, 7-vegetative state, 6-lower severe disability, 5-upper severe disability, 4-lower moderate disability, 3-upper moderate disability, 2-lower good recovery, 1-upper good recovery)
Pediatric Quality of Life Inventory (PedsQL) Multidimensional Fatigue Scale | 1 week, 1 month, 3 months, and 6 months
  Fatigue and cognitive function; 0 to 100 with higher scores representing better outcomes
D-dimer | Change from baseline to end of 8-hour study drug infusion
  Measure clot breakdown (ng/mL)
Plasmin-antiplasmin (PAP) complex | Change from baseline to end of 8-hour study drug infusion
  Measure fibrinolytic activity (mcg/L)
Tissue plasminogen activator (tPA) | Change from baseline to end of 8-hour study drug infusion
  Measure fibrinolytic activity (ng/mL)
Thrombosis | 1 week or at hospital discharge (whichever comes first)
  Any venous or arterial thrombosis on standard diagnostic imaging post-randomization
Seizure | 1 week or at hospital discharge (whichever comes first)
  Clinical or electroencephalogram-documented seizure
Behavior Rating Inventory of Executive Function (BRIEF) | 6 and 12 months after injury
  Measurement of executive function after traumatic brain injury

CONTACTS AND LOCATIONS:
Overall Officials: Daniel K Nishijima, MD, MAS, Principal Investigator — University of California, Davis; Nathan Kuppermann, MD, MPH, Principal Investigator — University of California, Davis

IPD SHARING:
Plan to Share IPD: Yes
A public use database will be produced and will be completely de-identiﬁed in accordance with the deﬁnitions provided in the Health Insurance Portability and Accountability Act (HIPAA).
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 12 months after publication of primary manuscript.
Access Criteria: Approval through NIH and PECARN
URL: https://pecarn.org/datasets/

REFERENCES:
- [Result] Nishijima DK, Gosdin M, Naz H, Tancredi DJ, Hewes HA, Myers SR, Stanley RM, Adelson PD, Burd RS, Finkelstein Y, VanBuren J, Casper TC, Kuppermann N; TIC-TOC Collaborators of the Pediatric Emergency Care Applied Research Network (PECARN). Assessment of primary outcome measures for a clinical trial of pediatric hemorrhagic injuries. Am J Emerg Med. 2021 May;43:210-216. doi: 10.1016/j.ajem.2020.03.001. Epub 2020 Mar 9. PMID 32278572
- [Result] Trappey AF 3rd, Thompson KM, Kuppermann N, Stephenson JT, Nuno MA, Hewes HA, Meyers SR, Stanley RM, Galante JM, Nishijima DK; Traumatic Injury Clinical Trial Evaluating Tranexamic Acid in Children (TIC-TOC) Collaborators of the Pediatric Emergency Care Applied Research Network (PECARN). Development of transfusion guidelines for injured children using a Modified Delphi Consensus Process. J Trauma Acute Care Surg. 2019 Oct;87(4):935-943. doi: 10.1097/TA.0000000000002432. PMID 31299040
- [Result] Powers PE, Shore KK, Perez S, Ritley D, Kuppermann N, Holmes JF, Tzimenatos LS, Shawargga H, Nishijima DK. Public Deliberation as a Novel Method for an Exception From Informed Consent Community Consultation. Acad Emerg Med. 2019 Oct;26(10):1158-1168. doi: 10.1111/acem.13827. Epub 2019 Jul 24. PMID 31271691
- See also: TIC-TOC trial website — https://tictoctrial.org/